CLINICAL TRIAL: NCT05270109
Title: Cold Steel Versus "Hot" BiZact Tonsillectomy; Comparing Post Tonsillectomy Morbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Line Schiøtt Nissen (Other)
Collaborators: Sygehus Lillebaelt (Other); Sonderborg Hospital (Other Government); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Line Schiøtt Nissen, MD, Regional Hospital West Jutland
Organization: Regional Hospital West Jutland (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2202151
Record Dates: First submitted 2022-02-15; First posted 2022-03-08 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Tonsillectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BiZact (Experimental)
  Interventions: Procedure: BiZact
- Cold Steel (Active Comparator)
  Interventions: Procedure: Cold Steel

INTERVENTIONS:
Procedure: BiZact — In the "hot group" the peritonsillar space is dissected and sealed in one step by a bipolar instrument (BiZactTM). The instrument uses Valley Lab adjustable bipolar energy. Energy is automatically adjusted and delivered to the tissue in order minimize thermal tissue damage and seal blood vessels less than 3mm in diameter while dividing the soft tissue.
  Arms: BiZact
Procedure: Cold Steel — In the "cold steel group" the peritonsillar space is dissected with metal instruments, and bleeding is typically controlled by ligation or electrocautery.
  Arms: Cold Steel

SUMMARY:
Tonsillectomy, with or without adenoidectomy, in both children and adults is worldwide one of the most commonly performed surgical procedures in otorhinolaryngology, and the number is increasing. Alone in Denmark, approximately 8.000 tonsillectomies are performed annually. Although, tonsillectomy on benign indication is considered to be a minor and frequently performed surgical procedure, the operation is associated with significant morbidity. Postoperative pain and post tonsillectomy haemorrhage (PTH) are the most frequent, and PTH is potentially life threatening. In cold steel tonsillectomy, the peritonsillar space is dissected with metal instruments, and bleeding is typically controlled by ligation or electrocautery. This method has been used for the past 50 years, and is considered the "Gold Standard". However, new so-called "hot techniques have been developed. One of these is an impedance-dependent tissue sealer device (BiZactTM). The equipment used for BiZactTM tonsillectomy is EC certificated (CE nr. 00500). The equipment is commonly used for tonsillectomy both internationally and in Denmark, and preliminary results in both adults and children are promising. However, when a gold standard technique is replaced by a new technique, it is recommended that the decision is based on evidence obtained in randomized controlled designs, and preferably as a multicenter study.

Within the scope of the CE marking of the equipment, the purpose of the present study is to conduct a randomized controlled trial (RCT) in order to investigate whether tonsillectomy performed with BiZactTM "hot" technique is beneficial or at least non-inferior compared to the gold standard cold steel technique in terms of affecting the incidence of post-tonsillectomy morbidity, interoperative factors, patient satisfaction, and health related quality of life.

DETAILED DESCRIPTION:
Tonsillectomy, with or without adenoidectomy, conducted in both children and adults is worldwide one of the most commonly performed surgical procedures in otorhinolaryngology, and the number of tonsillectomies has increased over the recent decades. In Denmark, approximately 8.000 tonsillectomies are performed annually. The main indications for surgery are recurrent episodes of acute tonsillitis or upper airway obstruction due to adenotonsillar hypertrophy.

Although commonly performed, tonsillectomy is associated with significant morbidity of which postoperative pain and post tonsillectomy haemorrhage (PTH) are the most frequent. PTH is a major and potentially life-threatening complication of tonsil surgery. Postoperative pain lasts for approximately two weeks, and may in severe cases result in delayed discharge, a visit at the emergency department or readmission for pain control, re-hydration, and treatment of possible underlaying infection. The incidences of PTH vary between 0.3 and more than 10%. This variation may be caused by different definitions of PTH, but also differences in populations and indications. Cold steel tonsillectomy is considered to be the gold standard surgical technique, but several hot techniques including bipolar techniques, diathermy, and coblation have been developed and used for tonsillectomy. Until now these hot instruments have not proven better than the gold standard technique in reducing PTH, and it is recommended, that these hot techniques should be used with caution. Recently, a new Impedance-dependent tissue sealer device (BiZactTM) has been manufactured and approved for tonsil operations (19). Preliminary results are promising in terms of a PTH rate of 4.5%, a shortened operative time in the hands of both experienced and training surgeons with a median time of 5.1 minutes (range 1.5-26.5 minutes), and a reduced intraoperative blood loss between 1-10 milliliters.

Ideally, when a gold standard technique is replaced by a new technique, it is recommended that the decision should be based on evidence provided by RCTs involving several centers.

The aim of the present is to conduct a RCT to investigate whether tonsillectomy performed with a new hot technique (BiZactTM) is beneficial or at least non-inferior to the gold standard cold steel technique in terms of incidence of post-tonsillectomy morbidity, interoperative factors, patient satisfaction, and health related quality of life.

The study design is a double blind, multi-centre randomised controlled trial (RCT).

Patients, assessors, and investigators will be blinded to randomisation outcome.

Patients will be recruited at five Dept. Otorhinolaryngology: Region Hospital West, Holstebro, DK, Southwest Regional Hospital, Esbjerg, DK, Lillebaelt Regional Hospital, Vejle, DK, Southern Regional Hospital, Soenderborg, DK, and Aalborg University Hospital, Aalborg, DK.

A total of 1250 eligible patients referred to tonsillectomy on benign indication, who fulfil inclusion criteria and have signed declaration of consent, will be enrolled and randomised in the study; 625 patients are randomized to surgery performed by steel devices (Cold steel group), and 625 patients to surgery by an electrosurgical device (BiZactTM) (Hot group)

In the "cold steel group" the peritonsillar space is dissected with metal instruments, and bleeding is typically controlled by ligation or electrocautery. In the "hot group" the peritonsillar space is dissected and sealed in one step by a bipolar instrument (BiZactTM). The instrument uses Valley Lab adjustable bipolar energy. Energy is automatically adjusted and delivered to the tissue in order minimize thermal tissue damage and seal blood vessels less than 3mm in diameter while dividing the soft tissue.

An Inter-Rim analysis will be conducted after 650 included patients have fulfilled the study protocol.

In order to strengthen study homogeneity, a pilot-study will initially be carried out with the first ten patients at each of the involved otorhinolaryngology departments.

Randomization is computer generated. Random sequences of 5000 numbers with equal numbers of group assignments will be obtained and concealed at the Tonsil database website (www.tonsil.dk).

Randomisation will be performed automatically by ticking a box on a page of the Tonsil database website.

At the preoperative consultation or at the emergency department, a doctor not involved in the study, will establish registration of the patient in the database and carry out the randomisation.

After the randomisation procedure has been carried out, the outcome will be registered on a hidden page of the Tonsil database website, and it will not be possible to change the outcome. The randomization outcome will only be visible on the web-page from the day of surgery to the day after surgery. Hereafter, it will not be possible to see the randomisation outcome. The operating surgeon will not be able to influence the randomisation outcome.

The investigators hypothesise, that tonsillectomy performed with a bipolar electrosurgical device (BiZactTM) is noninferior to tonsillectomy performed with cold steel technique in terms of affecting postoperative morbidity defined as PTH demanding reoperation with haemostasis and pain.

The present study will elucidate whether tonsillectomy performed with a bipolar electrosurgical instrument BiZactTM induces alleged beneficial effects or at least is noninferior to tonsillectomy performed with cold steel instruments. Moreover, should the study uncover that tonsillectomy performed with a bipolar electrosurgical instrument BiZactTM can reduce postoperative morbidity, frequency of reoperations, as well as surgical time, it may potentially optimise future treatment for patients and reduce socio-economic costs. Thus, the present RCT will be followed with an alongside economic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Obstruction/ tonsillar hypertrophy.
* Recurrent tonsillitis, including previous peritonsillar abscess
* Chronic tonsillitis
* Systemic complications to tonsillitis (glomerulonephritis)
* Other (Mononucleosis), PFAPA (Periodic Fever, Aphtous stomatitis, pharyngitis, cervical adenitis)
* Foetor ex ore (tonsillar plugs)
* Peritonsillar abscess (Tonsillectomy a chaud)
* Ability to understand the written patient information and to give informed consent

Exclusion Criteria:

* Diseases in the hematopoietic system
* Antithrombotic or anticoagulant drugs in the recovery period
* Suspicion of/known tonsillar malignancies or other malignancy
* Patients or caregivers unable to read or speak Danish
* Patients or caregivers unable to use online application for self-evaluation

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Incidence of PTH | 24 hours until 30 days after surgery
  • Incidence of PTH defined as haemorrhage requiring haemostasis with; bipolar electric coagulation, ligature, compression and/or medical treatment with antifibrinolyticum within the first 24 hours after surgery until 30 days after surgery.
Postoperative pain | From the day of surgery until 14 days after the surgery
  • Postoperative pain assessed on a 11point numeric rating scale ranging from 0 "no pain" to 10 "worst possible pain". The Wong-Baker Faces rating scale is used for children.

SECONDARY OUTCOMES:
Blood loss | Intraoperative
  • Intraoperative blood loss assessed by standardized blood weighing. The weight in grams will be converted to milliliters.
Knife time | First day of surgery
  • Operative time in minutes from the Boyle-Davis gag is placed until it is removed.
PROM | From the day of the surgery until 6 months after the surgery
  • patient reported outcome measures (PROM) of postoperative recovery (days until return to normal diet, days until return to physical activity, and days until return to work, school- or child care).
Unscheduled contacts to the health care system | From the day of the surgery until 14 days after
  - Number of unscheduled contacts to the health care system.
Health related quality of life | From the day of the surgery until 6 months after the surgery
  • Health related quality of life using EQ5D
Smell and taste | From the day of the surgery until 6 months after the surgery
  Smell and taste validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Line S Nissen, MD, Principal Investigator — Regional Hospital West Jutland
Locations (1):
- Line Schiøtt Nissen, Gødstrup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molhave M, Lyhne NM, Jensen DF, Nielsen SH, Hahn P, Holm JK, Ovesen T, Bertelsen J. BiZact versus cold steel for post-tonsillectomy hemorrhage: a multicenter randomized trial. Eur Arch Otorhinolaryngol. 2025 Dec;282(12):6449-6457. doi: 10.1007/s00405-025-09703-3. Epub 2025 Oct 13. PMID 41083818
- [Derived] Nissen LS, Bertelsen J, Lyhne NM, Nielsen SH, Hahn P, Holm J, Ovesen T. Cold steel versus impedance-dependent tissue sealer tonsillectomy - a study protocol for a randomised controlled trial. Dan Med J. 2023 Nov 23;70(12):A06230366. PMID 38018707